CLINICAL TRIAL: NCT03428659
Title: Dynamic Time Series Data Collection for Functional Recovery Changes in Sub-acute Stroke Patients
Brief Title: Functional Recovery Changes in Subacute Stroke Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-11-081
Record Dates: First submitted 2018-02-04; First posted 2018-02-09 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2019-09

CONDITIONS: Sub-acute Stroke
Keywords: Motor function; Recovery; Gait; Magnetic resonance imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sub-acute stroke: More than 1 week post-stroke Ischemic or hemorrhagic stroke
  Interventions: Other: Data acquisition of functional abilities in sub-acute stroke

INTERVENTIONS:
Other: Data acquisition of functional abilities in sub-acute stroke — MRI data, motor evoked potentials, gait function and behavior data acquisition

SUMMARY:
In subacute stroke patients, dynamic time series data of brain imaging and motor function measurement were obtained from 7 days to 6 months (total 9 times) after stroke onset

ELIGIBILITY:
Inclusion Criteria:

* at least 19 years of age hemiplegic stroke patients
* Subacute-phase ischemic or hemorrhagic stroke patients within 7 days of onset
* Functional Ambulation Category Scale (FAC) of 3 or less, 7 days of onset,
* A person who understands and voluntarily participates in this study and signs a research agreement

Exclusion Criteria:

* User of artificial heartbeat
* Patients with claustrophobia
* Patients with metal implants
* Patients who are contraindicated for other common MRI
* Patients with mild motor impairment with an FMA score of 80 or higher
* Patients whose conscious state is coma and who have no response at all
* Patients who can not independently gait with the Modified Rankin Scale (mRS) score of 4 or more before the onset of disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A person who was inpatient at sub-acute stage at the Samsung Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mechanism of recovery of motor function according to recovery of sub-acute stroke | Through study completion, an average of 6 months
  Mechanism of recovery of motor function calculate by repeated measurement method in physical and cognitive functions data and MRI data of brain
Mechanism of recovery of gait function according to recovery of sub-acute stroke | Through study completion, an average of 6 months
  Mechanism of recovery of motor function calculate by repeated measurement method in 3D motion capture system and electromyography (EMG) data and MRI data of brain

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No